CLINICAL TRIAL: NCT04338620
Title: An Explorative Study on Camrelizumab Combined With Albumin-bound Paclitaxel and Platinum in Neoadjuvant Treatment of Resectable Non-small-cell Lung Carcinoma
Brief Title: Camrelizumab Combined With Albumin-bound Paclitaxel and Platinum in Neoadjuvant Treatment of Resectable NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XBSX-L1-002
Record Dates: First submitted 2020-04-06; First posted 2020-04-08 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Non-small-cell Lung Cancer (NSCLC)
Keywords: Camrelizumab; neoadjuvant treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Platinum; Albumin-Bound Paclitaxel

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, open-label, parallel controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Experimental Group (Experimental): Participants receive totally 3 cycles of camrelizumab combined with albumin-bound paclitaxel and Cisplatin/carboplatin/Nedaplatin treatment during preoperative period, every 3 weeks for up to 3 cycles.
  Interventions: Drug: camrelizumab、albumin-bound paclitaxel and platinum
- B: Control group (Active Comparator): Participants receive totally 3 cycles of albumin-bound paclitaxel combined with Cisplatin/carboplatin/Nedaplatin treatment during preoperative period, every 3 weeks for up to 3 cycles.
  Interventions: Drug: albumin-bound paclitaxel and platinum

INTERVENTIONS:
Drug: camrelizumab、albumin-bound paclitaxel and platinum — Experimental Group：camrelizumab、albumin-bound paclitaxel and platinum. Camrelizumab will be administered as a 30-minute IV infusion Q3W at a dose of 200mg on day1 of each cycle. Albumin-bound paclitaxel will be administered as a 30-minute IV infusion Q3W at a dose of 130 mg/m2 on day1 and day8 of each cycle. Platinum included Cisplatin/carboplatin/Nedaplatin
  Arms: A: Experimental Group
Drug: albumin-bound paclitaxel and platinum — Control group：albumin-bound paclitaxel and platinum. Albumin-bound paclitaxel will be administered as a 30-minute IV infusion Q3W at a dose of 130 mg/m2 on day1 and day8 of each cycle.
  Platinum included Cisplatin/carboplatin/Nedaplatin
  Arms: B: Control group

SUMMARY:
Explorative study, which evaluates the effect of Camrelizumab combined with albumin-bound paclitaxel and platinum in neoadjuvant treatment of resectable non-small-cell lung carcinoma.

DETAILED DESCRIPTION:
This is a multicenter, randomized, open parallel controlled trial to evaluate the efficacy and safety of camrelizumab combined with albumin-bound paclitaxel and platinum versus albumin-bound paclitaxel combined with platinum in resectable stage IIIA -IIIB NSCLC (IIIB is limited toT3N2).

ELIGIBILITY:
Inclusion Criteria:

* Age :18 Years to 70 Years (Adult, Older Adult)
* ECOG physical score status of 0 or 1 points;
* expected survival time ≥ 12 weeks;
* Pathological diagnosis with StageIIIA-IIIB NSCLC;
* According to the eighth edition of the AJCC/UICC TNM staging system, patients was pathological diagnosed with Stage III-N2 clinically resectable NSCLC.
* Patients with at least one evaluable or measurable lesions as per RECIST version 1.1 （CT scan length and diameter of tumor lesion≥10mm，CT scan of lymph node lesion was short diameter≥15mm；）
* Patients were newly diagnosed with non-small cell lung cancer, without radiotherapy, chemotherapy, surgery or molecule-targeted treatment.
* Patients must have enough cardiopulmonary function for the expected pulmonary resections for lung cancer.
* The main organ function meets the following criteria:1) blood routine:a. ANC ≥ 1.5×109/L; b. PLT ≥ 100×109/L; c. HB ≥ 90 g/L; 2) Blood biochemistry:TBIL ≤ 1.5×ULN;ALT、AST≤ 2.5×ULN;sCr≤1.5×ULN; 3) Blood coagulation: INR≤1.5×ULN and APTT≤1.5×ULN，endogenous creatinine clearance rate≥50ml/min(Cockcroft-Gault formula);
* Pregnancy test (serum or urine) has to be performed for woman of childbearing age within 7 days before enrolment and the test result must be negative. They shall take appropriate methods for contraception during the study until the 3 months post the last administration of study drug. For men, (previous surgical sterilization accepted), shall agree to take appropriate methods of contraception during the study until the 3 months post the last administration of study drug;
* Patient has to voluntarily join the study and sign the Informed Consent Form for the study.

Exclusion Criteria:The subject must be excluded from participating in the trial if the subject:

* Patients with brain metastasis
* Patients with autoimmune disease, or a history of autoimmune disease including but not limited to the following: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism which can be included after hormone replacement therapy; Subjects with childhood asthma have been completely alleviated and without any intervention or vitiligo in adulthood can be included.
* Subjects who need medical intervention with bronchodilators cannot be included.
* Subjects with congenital or acquired immunodeficiency such as HIV infection, active hepatitis B (HBV DNA ≥ 2000 IU/mL), hepatitis C (hepatitis C antibody is positive);
* Subjects with a condition requiring other immunosuppressive medications before 14 days of study drug administration firstly, not including inhaled corticosteroids or physiological doses of systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents).
* Has received a live vaccine within 4 weeks of planned start of study therapy.
* Other malignancies have been diagnosed within 3 years prior to the first use of the study drug; 8. Patients with a current or history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiologic pneumonia, drug-induced pneumonia and severe impairment of lung function.
* Patients with hypertension that is difficult to control (systolic blood pressure ≥140 mmHg and diastolic blood pressure ≥90 mmHg);
* patients with myocardial ischemia and myocardial infarction above class II (including QT interval prolongation, for man ≥ 450 ms, for woman ≥ 470 ms);
* Severe infection within 4 weeks before the first administration (such as intravenous drip of antibiotics, antifungal drugs or antiviral drugs), or fever of unknown origin (> 38.5 ℃) within 4 weeks before the first administration.
* allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation.
* Pregnant or nursing women; 14. Patients with a history of hypersensitivity to any of the study drugs, similar drugs, or excipients.
* Participated in other clinical trials within 4 weeks; 16. Patients with the history of drug abused or alcohol.
* The investigator believes that there are any conditions that may damage the subject or result in the subject being unable to meet or perform the research request;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2020-04-07 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
pathological complete response (pCR) | The day of the surgery
  no residual tumor cells in the surgically resected tumor specimen and all sampled regional lymph nodes after neoadjuvant treatment.

SECONDARY OUTCOMES:
main pathology rate (MPR) | The day of the surgery
  Major pathological response rate (MPR): defined as ≤ 10% of residual tumor cells in the surgically resected tumor specimen and sampled regional lymph nodes after neoadjuvant treatment.
Objective Response Rate (ORR) | pre-operation
  Objective response rate (ORR): defined as the proportion of patients whose tumor size shrinks to predefined values，which including cases of CR and PR. Objective tumor response will be assessed using RECIST 1.1. Subjects must have measurable tumor lesions at baseline, and the response evaluation criteria are classified as complete response (CR), partial response (PR), stable disease (SD), and progressive disease (PD) according to RECIST 1.1.
Event-free Survival （EFS） | Event-free survival (EFS): defined as the time from the randomization until the date of first documented progression or recurrence or date of death from any cause, whichever came first, assessed up to 100 months
  Event-free survival (EFS): defined as the time from the randomization to the first occurrence of disease progression or recurrence, or death (due to any cause).
Assess adverse events | 90 days
  Assess all adverse events according to the NCI Common Terminology Criteria for (NCI CTCAE) v5.

OTHER OUTCOMES:
type of surgery、R0 Resection、Surgical approach、Duration from final treatment to surgery、Duration of surgery、Length of hospital stay and rate of peri- and post-operative complications | within 30 days of surgery
  enumeration data：type of surgery、R0 Resection、Surgical approach
  measurement data：Duration from final treatment to surgery、Duration of surgery、Length of hospital stay.
  Peri- and post-operative complications reported up to 30 days after surgery. The Clavien-Dindo scale classifies peri- and post-operative complications into 5 grades.complications (within 30 days of surgery) in subjects treated with camrelizumab plus chemotherapy compared to those treated with chemotherapy alone.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Tao, PhD, Principal Investigator — The Fourth Military Medical University Tangdu Hospital
Locations (1):
- The Fourth Military Medical University Tangdu Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lei J, Zhao J, Gong L, Ni Y, Zhou Y, Tian F, Liu H, Gu Z, Huang L, Lu Q, Wang X, Sun J, Yang E, Wang T, Zhong D, Wang J, Zhao Z, Liu Z, Wang C, Wang X, Lei G, Yan X, Jiang T. Neoadjuvant Camrelizumab Plus Platinum-Based Chemotherapy vs Chemotherapy Alone for Chinese Patients With Resectable Stage IIIA or IIIB (T3N2) Non-Small Cell Lung Cancer: The TD-FOREKNOW Randomized Clinical Trial. JAMA Oncol. 2023 Oct 1;9(10):1348-1355. doi: 10.1001/jamaoncol.2023.2751. PMID 37535377